CLINICAL TRIAL: NCT04438811
Title: Task-based Credentialing for Medical Officers in Spinal Anesthesia: An Innovative Approach to the Specialist Workforce Crisis in Rural Indian Hospitals Curriculum Training of Medical Officers
Brief Title: Task-based Credentialing for Medical Officers in Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Ashwini Health System, Gudalur, India (Unknown); Harvard Center for Global Health, Dubai (Unknown); Boston Children's Hospital (Other); Program in Global Surgery and Social Change, Harvard Medical School (Unknown)
Responsible Party: Principal Investigator, Craig McClain, Principle Investigator, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0624
Record Dates: First submitted 2020-06-08; First posted 2020-06-19 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Spinal Anesthesia; Task Sharing in Anesthetic Delivery in Areas With Limited Access to Care
Keywords: global health

STUDY DESIGN:
Intervention Model Description: This is a non-inferiority, randomized trial. Patients will be randomized to receive a protocolized spinal anesthetic from a consultant anesthetist or a trained medical officer. Failure rates and need for rescue will be assessed as primary outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consultant Anesthetist (Other): Patients who are randomized to this arm will receive their spinal anesthesia froma consultant anesthetist
  Interventions: Other: delivery of spinal anesthetic by a consultant anesthetist
- Medical Officer (Other): Patients randomized to this arm will receive their spinal anesthetic from a medical officer. There will be a consultant anesthetist immediately available if needed but they will not be a direct participant in this arm. Any involvement by the consultant will result in the label of failure for this patient.
  Interventions: Other: delivery of the spinal anesthetic by a trained medical officer

INTERVENTIONS:
Other: delivery of the spinal anesthetic by a trained medical officer — The delivery of spinal anesthesia by the trained medical officers in 3 rural Indian hospitals will be compared to those delivered by consultant anesthetists in the same hospitals in a non-inferiority analysis.
  Arms: Medical Officer
Other: delivery of spinal anesthetic by a consultant anesthetist — The delivery of spinal anesthesia by the trained medical officers in 3 rural Indian hospitals will be compared to those delivered by consultant anesthetists in the same hospitals in a non-inferiority analysis.
  Arms: Consultant Anesthetist

SUMMARY:
Test the safety and effectiveness of training medical officers in the provision of spinal anesthesia in a rural hospital context using a non-inferiority randomized trial.

The safety and effectiveness of the MOs will be evaluated through a non-inferiority trial in which patients are randomized to care by a trained MO or an anesthesiologist. The primary outcomes are safety (adherence to adapted anesthesia safety checklist- see supporting documents "Adapted Anesthesia Safety Checklist") and effectiveness (adequate analgesia) of spinal anesthesia.

DETAILED DESCRIPTION:
The vast majority of the world is without access to surgical and anesthesia care, and a severe workforce shortage is a major contributing factor. The Lancet Commission on Global Surgery (LCoGS) demonstrated that Africa and South Asia, home to over a third of the global population, lay claim to just 12% of surgeons, anesthesiologists and obstetricians. This workforce shortage may be particularly severe for anesthesia care given that anesthesiologist make up less than 20% of surgical care providers globally. In a series of qualitative interviews, providers across three continents noted that in rural and under-resourced areas, it was unlikely that there was a surgeon and an anesthesiologist in the same place.

In India, the concerns of under-provision of human resources in the rural area are especially severe. The Lancet commission on Global Surgery estimates that while 68% of Indians live in rural areas, only 22% of the health care workforce does. For specialist services, which are even more urbanized, the disparity is likely greater. The result is that, in South Asia, 95% of people are estimated to lack access to safe, affordable and timely surgical care.

In India, which is home to nearly 400 medical schools, it may be posited that the country is well positioned to close this gap. However, the number of postgraduate training seats - 14,000 countrywide - are entirely insufficient for the 50,000 doctors that graduate each year. With only 1500 postgraduate training seats for anesthesia, a graduate who may otherwise aspire to train in anesthesia instead remains generalist MO or seeks training elsewhere. The World Health Organization suggests that a presence of anesthesiologists in rural India may be so scarce it is "non-existent.". It has also been estimated that 43% of the Indian population lives more than 50km from their nearest health center, 76% of which do not have an anesthesiologist.

The result of these human resource limitations, is that rural Indian surgeons often administer anesthesia for their patient prior to performing necessary surgeries or medical officers with only ad hoc training provide anesthesia care. The de facto standard of care in rural India, ends up being the provision of anesthesia by a surgeon or untrained medical officer. While advocacy towards increasing post-graduate education must continue, it is also clear that interim measures are needed to improve upon current baseline practices.

One such measure suggested by the Disease Control Priorities 3 (DCP3), the LCoGS, and others is the concept of "task-based credentialing." In this model of credentialing, physicians are trained and credentialed in a limited set of procedures. Task sharing - a process by which non-specialists take on whole-sale the tasks typically performed by a specialist - is prevalent in the provision of anesthesia care worldwide. However, a recent meta-analysis evaluated outcomes for task-sharing in anesthesia in 15 LMIC and found that administration of anesthesia by a non-physician was a risk-factor for maternal mortality. To mitigate these concerns, task-based credentialing focuses on the training of non-specialist medical officers in a discrete, well-defined task and includes training to deal with the possible complications. This task-based training would serve as an improvement on the de facto standard of care in rural India by providing specific training in place of ad hoc learning.

The provision of spinal anesthesia is thought to be well-suited for this form of training. The procedure involves the injection of a local anesthetic agent into the subarachnoid space. This allows for analgesia and anesthesia below the level of injection. This procedure is widely used in general surgery, obstetric surgery, and orthopedic surgery. Moreover, the use of spinal anesthesia is particularly well-adapted to rural care as it is less expensive than general anesthesia and has a lower requirement of infrastructure and disposables when compared to general anesthesia.

Test the safety and effectiveness of training medical officers in the provision of spinal anesthesia in a rural hospital context using a non-inferiority randomized trial.

The safety and effectiveness of the MOs will be evaluated through a non-inferiority trial in which patients are randomized to care by a trained MO or an anesthesiologist. The primary outcomes are safety (adherence to adapted anesthesia safety checklist- see supporting documents "Adapted Anesthesia Safety Checklist") and effectiveness (adequate analgesia) of spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for MOs

* Consent to participate in practical training and clinical trial (consent process will be repeated)
* Successful completion of the theoretical and simulation training
* Be deemed safe to continue to practical training by their supervising Anesthesiologist
* Feel comfortable to proceed to practical training

Inclusion criteria for patients

* Age 18-65
* Undergoing one of the surgeries noted in supporting document "List of surgeries for patient inclusion criteria" or otherwise deemed appropriate for spinal anesthesia as determined by surgeon and supervising anesthesiologist

  * Willingness to provide informed consent
  * ASA (American Society of Anesthesiology Physical Status Classification System) grades I and II

Inclusion criteria for Consultant Anesthetists

* Anesthetist licensed to practice independently with availability to provide care at one of the selected sites

Exclusion Criteria:

Exclusion criteria for MOs

* Recent suspension from clinical practice
* Due to change sites or retire before the expected end date of the trial

Exclusion criteria for patients

* Obese (BMI > 35)
* Refusal of consent to participate in trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Successful delivery of spinal anaesthesia | Assessed pre-operatively following recruitment and consent (day 0 of the follow up period)
  Delivery of spinal anaesthesia into the intrathecal space with three or less attempts and no intra-operative conversion to general anaesthesia due to spinal failure

SECONDARY OUTCOMES:
Post-operative Complications | Reviewed at two time points - on discharge from healthcare facility or day 3 post-operatively (whichever occurs first) and day 10-14 post-operatively
  Incidence of post-dural puncture headache, epidural haematoma, spinal abscess and neurological deficit
Patient experience measures | Reviewed at two time points - on discharge from healthcare facility or day 3 post-operatively (whichever occurs first) and day 10-14 post-operatively
  Patient reported experience measures of clinical care and pain
Intraoperative Complications | Assessed intraoperatively during surgical procedure
  The incidence of hypotension, bradycardia, high spinal, apnoea and hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Craig D McClain, MD, MPH, Principal Investigator — Boston Children's Hospital, Harvard Medical School, Program in Global Surgery and Social Change
Locations (4):
- Boston Children's Hospital, Boston, Massachusetts, United States
- India (3):
  - JSS Hospital, Ganiyari, Chhattisgarh
  - Ashwini Hospital, Gudalur, Tamil Nadu
  - Sittilingi Tribal Hospital, Harūr, Tamil Nadu

REFERENCES:
- [Background] Meara JG, Leather AJ, Hagander L, Alkire BC, Alonso N, Ameh EA, Bickler SW, Conteh L, Dare AJ, Davies J, Merisier ED, El-Halabi S, Farmer PE, Gawande A, Gillies R, Greenberg SL, Grimes CE, Gruen RL, Ismail EA, Kamara TB, Lavy C, Lundeg G, Mkandawire NC, Raykar NP, Riesel JN, Rodas E, Rose J, Roy N, Shrime MG, Sullivan R, Verguet S, Watters D, Weiser TG, Wilson IH, Yamey G, Yip W. Global Surgery 2030: evidence and solutions for achieving health, welfare, and economic development. Lancet. 2015 Aug 8;386(9993):569-624. doi: 10.1016/S0140-6736(15)60160-X. Epub 2015 Apr 26. No abstract available. PMID 25924834
- [Background] Grimes CE, Bowman KG, Dodgion CM, Lavy CB. Systematic review of barriers to surgical care in low-income and middle-income countries. World J Surg. 2011 May;35(5):941-50. doi: 10.1007/s00268-011-1010-1. PMID 21360305
- [Background] Hoyler M, Finlayson SR, McClain CD, Meara JG, Hagander L. Shortage of doctors, shortage of data: a review of the global surgery, obstetrics, and anesthesia workforce literature. World J Surg. 2014 Feb;38(2):269-80. doi: 10.1007/s00268-013-2324-y. PMID 24218153
- [Background] Bergstrom S, McPake B, Pereira C, Dovlo D. Workforce Innovations to Expand the Capacity for Surgical Services. In: Debas HT, Donkor P, Gawande A, Jamison DT, Kruk ME, Mock CN, editors. Essential Surgery: Disease Control Priorities, Third Edition (Volume 1). Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2015 Apr 2. Chapter 17. Available from http://www.ncbi.nlm.nih.gov/books/NBK333504/ PMID 26741003
- [Background] Holmer H, Lantz A, Kunjumen T, Finlayson S, Hoyler M, Siyam A, Montenegro H, Kelley ET, Campbell J, Cherian MN, Hagander L. Global distribution of surgeons, anaesthesiologists, and obstetricians. Lancet Glob Health. 2015 Apr 27;3 Suppl 2:S9-11. doi: 10.1016/S2214-109X(14)70349-3. No abstract available. PMID 25926323
- [Background] Dubowitz G, Detlefs S, McQueen KA. Global anesthesia workforce crisis: a preliminary survey revealing shortages contributing to undesirable outcomes and unsafe practices. World J Surg. 2010 Mar;34(3):438-44. doi: 10.1007/s00268-009-0229-6. PMID 19795163
- [Background] Ng-Kamstra JS, Greenberg SLM, Abdullah F, Amado V, Anderson GA, Cossa M, Costas-Chavarri A, Davies J, Debas HT, Dyer GSM, Erdene S, Farmer PE, Gaumnitz A, Hagander L, Haider A, Leather AJM, Lin Y, Marten R, Marvin JT, McClain CD, Meara JG, Mehes M, Mock C, Mukhopadhyay S, Orgoi S, Prestero T, Price RR, Raykar NP, Riesel JN, Riviello R, Rudy SM, Saluja S, Sullivan R, Tarpley JL, Taylor RH, Telemaque LF, Toma G, Varghese A, Walker M, Yamey G, Shrime MG. Global Surgery 2030: a roadmap for high income country actors. BMJ Glob Health. 2016 Apr 6;1(1):e000011. doi: 10.1136/bmjgh-2015-000011. eCollection 2016. PMID 28588908
- [Background] Raykar NP, Yorlets RR, Liu C, Greenberg SL, Kotagal M, Goldman R, Roy N, Meara JG, Gillies RD. A qualitative study exploring contextual challenges to surgical care provision in 21 LMICs. Lancet. 2015 Apr 27;385 Suppl 2(Suppl 2):S15. doi: 10.1016/S0140-6736(15)60810-8. Epub 2015 Apr 26. PMID 26313061
- [Background] Alkire BC, Raykar NP, Shrime MG, Weiser TG, Bickler SW, Rose JA, Nutt CT, Greenberg SL, Kotagal M, Riesel JN, Esquivel M, Uribe-Leitz T, Molina G, Roy N, Meara JG, Farmer PE. Global access to surgical care: a modelling study. Lancet Glob Health. 2015 Jun;3(6):e316-23. doi: 10.1016/S2214-109X(15)70115-4. Epub 2015 Apr 27. PMID 25926087
- [Background] MUZAFFARNAGAR, I. Special Report: Why India's medical schools are plagued with fraud. Available from: http://www.reuters.com/article/us-india-medicine-education- specialrepor-idUSKBN0OW1NM20150617.
- [Background] Shetty, D., Reform medical education, transform healthcare, in The Times of India. 2015.
- [Background] Cherian M, Choo S, Wilson I, Noel L, Sheikh M, Dayrit M, Groth S. Building and retaining the neglected anaesthesia health workforce: is it crucial for health systems strengthening through primary health care? Bull World Health Organ. 2010 Aug 1;88(8):637-9. doi: 10.2471/BLT.09.072371. Epub 2010 May 10. No abstract available. PMID 20680130
- [Background] Dare AJ, Ng-Kamstra JS, Patra J, Fu SH, Rodriguez PS, Hsiao M, Jotkar RM, Thakur JS, Sheth J, Jha P; Million Death Study Collaborators. Deaths from acute abdominal conditions and geographical access to surgical care in India: a nationally representative spatial analysis. Lancet Glob Health. 2015 Oct;3(10):e646-53. doi: 10.1016/S2214-109X(15)00079-0. Epub 2015 Aug 13. PMID 26278186
- [Background] Jamison DT, Alwan A, Mock CN, Nugent R, Watkins D, Adeyi O, Anand S, Atun R, Bertozzi S, Bhutta Z, Binagwaho A, Black R, Blecher M, Bloom BR, Brouwer E, Bundy DAP, Chisholm D, Cieza A, Cullen M, Danforth K, de Silva N, Debas HT, Donkor P, Dua T, Fleming KA, Gallivan M, Garcia PJ, Gawande A, Gaziano T, Gelband H, Glass R, Glassman A, Gray G, Habte D, Holmes KK, Horton S, Hutton G, Jha P, Knaul FM, Kobusingye O, Krakauer EL, Kruk ME, Lachmann P, Laxminarayan R, Levin C, Looi LM, Madhav N, Mahmoud A, Mbanya JC, Measham A, Medina-Mora ME, Medlin C, Mills A, Mills JA, Montoya J, Norheim O, Olson Z, Omokhodion F, Oppenheim B, Ord T, Patel V, Patton GC, Peabody J, Prabhakaran D, Qi J, Reynolds T, Ruacan S, Sankaranarayanan R, Sepulveda J, Skolnik R, Smith KR, Temmerman M, Tollman S, Verguet S, Walker DG, Walker N, Wu Y, Zhao K. Universal health coverage and intersectoral action for health: key messages from Disease Control Priorities, 3rd edition. Lancet. 2018 Mar 17;391(10125):1108-1120. doi: 10.1016/S0140-6736(17)32906-9. Epub 2017 Nov 25. PMID 29179954
- [Background] Gnanaraj J, Jason LY, Khiangte H. High quality surgical care at low cost: the diagnostic camp model of Burrows Memorial Christian Hospital (BMCH). Indian J Surg. 2007 Dec;69(6):243-7. doi: 10.1007/s12262-007-0034-0. Epub 2008 Jan 28. PMID 23132995
- [Background] Federspiel F, Mukhopadhyay S, Milsom P, Scott JW, Riesel JN, Meara JG. Global surgical and anaesthetic task shifting: a systematic literature review and survey. Lancet. 2015 Apr 27;385 Suppl 2:S46. doi: 10.1016/S0140-6736(15)60841-8. Epub 2015 Apr 26. PMID 26313095
- [Background] Sobhy S, Zamora J, Dharmarajah K, Arroyo-Manzano D, Wilson M, Navaratnarajah R, Coomarasamy A, Khan KS, Thangaratinam S. Anaesthesia-related maternal mortality in low-income and middle-income countries: a systematic review and meta-analysis. Lancet Glob Health. 2016 May;4(5):e320-7. doi: 10.1016/S2214-109X(16)30003-1. PMID 27102195
- [Derived] Menon N, George R, Kataria R, Manoharan R, Brooks MB, Pendleton A, Sheshadri V, Chatterjee S, Rajaleelan W, Krishnan J, Sandler S, Saluja S, Ljungman D, Raykar N, Svensson E, Wasserman I, Zorigtbaatar A, Jesudian G, Afshar S, Meara JG, Peters AW, McClain CD. Task-sharing spinal anaesthesia care in three rural Indian hospitals: a non-inferiority randomised controlled clinical trial. BMJ Glob Health. 2024 Aug 16;9(8):e014170. doi: 10.1136/bmjgh-2023-014170. PMID 39153752